CLINICAL TRIAL: NCT06525233
Title: Comparision the Effect of Interval Aerobic Training and Continious Training on Coronary Artery Disease
Brief Title: Interval Aerobic Training and Continious Training
Status: Completed | Type: Observational
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, gulay karacaoglu, Dr., Istanbul Medipol University Hospital
Other Study IDs: aerobicexercise
Record Dates: First submitted 2019-08-17; First posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Coronary Artery Disease; Exercise Addiction
Keywords: continious training; interval training
MeSH Terms: conditions — Coronary Artery Disease | interventions — Physical Therapy Modalities; Rehabilitation

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Treatment: humans that diagnosed as coronary artery disease, joined two aerobic exercise groups. One of this group includes interval exercise and the other one includes continuous exercise.
  Interventions: Other: Physiotherapy and rehabilitation

INTERVENTIONS:
Other: Physiotherapy and rehabilitation — The aerobic exercise is very crucial part of cardiac rehabilitation. This study compares the effects of interval and continuous training which are the two types of aerobic training on persons' life quality and exercise capacity diagnosed coronary artery disease patients.

SUMMARY:
This research is comparing the effects of interval and continuous training which are the two types of aerobic training on persons' life quality and exercise capacity on coronary artery disease patients.

DETAILED DESCRIPTION:
The participants are diagnosed coronary artery disease aged between 40- 80 and have no mental and physical disability to take part in research. The participants' demographic infos and clinical story were recorded. To evaluate exercise capacity we used the symptom-limited exercise test (ETT) and six minute walking test (6DYT). We evaluate the life quality by using Short Form-36 (SF-36).

All those evaluation tests are done before and after training. Participants are randomly divided into two groups, the first group took part in interval aerobic training (AAE) while the other group was joining in continuous training (SAE) three times a week during 6 weeks. In both groups, significant changes were found in ETT, test time and 6 DYT scores after the rehabilitation program (p<0,05). But only AAE group have important statistical values comparing to SAE group on test time and 6DYT scores. After training SAE group showed significant statistical change in every SF-36 parameter, while AAE group showing significant values except energy/fatigue. AAE group have statistically significant changes comparing to SAE group on that parameters; physical function, role limitations due to physical function, role limitations due to emotional function and general health (p<0,05). Consequently AAE is much more tolerable comparing to SAE and AAE is considered more effective in increasing some parameters. On the other hand, we observed that both training types can be used in cardiac rehabilitation safely.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed coronary artery disease
* aged between 40-80
* over %55 ejection fraction

Exclusion Criteria:

* mental and physical disability
* unstable angina pectoris
* thrombophlebitis

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Name-Surname, age, sex, body-weight index, educational status, married/single/divorced, job and clinical background (If has any surgery and myocardial infarction)
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2018-05-05 (Actual); Primary Completion 2019-04-02 (Actual); Study Completion 2019-05-20 (Actual)

PRIMARY OUTCOMES:
the effect of intermittent and continuous aerobic exercise on exercise capacity | 30 minutes 3 times a week during 6 weeks
  we used the symptom-limited exercise test and six minute walking test (6DYT). All evaluation tests are done before and after training. Participants were into randomised two groups: interval aerobic training (AAE) and continuous aerobic training (SAE). Training lasted three times a week during 6 weeks. In both groups, significant changes were found in evaluation tests scores after the rehabilitation program (p<0,05). But only AAE group have important statistical difference comparing to SAE group on test time and 6DYT scores.

SECONDARY OUTCOMES:
the effect of intermittent and continuous aerobic exercise on life quality | 30 minutes 3 times a week during 6 weeks
  The participants have no mental and physical disability to join in research. The participants' demographic infos and clinical story were recorded.We evaluate the life quality by using Short Form-36 (SF-36). All evaluation tests are done before and after training. Participants were into randomised two groups: interval aerobic training (AAE) and continuous aerobic training (SAE).After training SAE group showed significant statistical change in every SF-36 parameter, while AAE group showing significant values except energy/fatigue. AAE group have statistically significant changes comparing to SAE group on that parameters; physical function, role limitations due to physical function, role limitations due to emotional function and general health (p<0,05). Consequently AAE is much more tolerable comparing to SAE and AAE is considered more effective in increasing some parameters. On the other hand, we observed that both training types can be used in cardiac rehabilitation safely.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Mutluay, Study Director — medipol univercity
Locations (1):
- Physiotherapy and Rehabilitation Center, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Cardiac rehabilitation is very popular at nowadays and which type exercise good on cardiac rehabilitation is not known exactly
Supporting Information: CSR
Time Frame: 2 years
Access Criteria: karacaoglugulay@gmail.com